CLINICAL TRIAL: NCT05998005
Title: Assessing Cultures of Recovery in Tribal Communities - Research Core - Training Evaluation
Brief Title: First Face Training Evaluation in Tribal Communities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Healing Lodge of the Seven Nations (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1S06GM146095-01-8249; 1S06GM146095 (NIH)
Record Dates: First submitted 2023-07-25; First posted 2023-08-18 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Mental Health; Substance-Related Disorders
Keywords: addiction; mental health; AI/AN; native american; american indian; mental health training program; training evaluation; NARCH; native american research centers for health; addictive behaviors; tribal participatory research; TPR
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Waitlist-control design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial training group (Experimental): Participants who are initially trained in the First Face training program
  Interventions: Behavioral: First Face Training Program
- Waitlist-control group (Other): Participants who are trained in the First Face training program 6 months after the initial training group
  Interventions: Behavioral: First Face Training Program

INTERVENTIONS:
Behavioral: First Face Training Program — First Face for Mental Health is a culturally-appropriate community-based mental health training for lay persons and others that prepares learners to provide assistance to someone having a mental health crisis. The course takes approximately 8 hours to complete.

SUMMARY:
The goal of this study is to evaluate a culturally grounded training curriculum, First Face for Mental Health, in Tribal communities, using a waitlist controlled trial design. This curriculum will train Tribal community members in how to respond to youth and adults experiencing mental health crises and serve as a bridge between these individuals and the help they need. The main questions the study aims to answer are:

* Does the training increase mental health knowledge, capacity and ability to respond to mental health situations, perceived competence to respond, and actual responsive actions among trainees?
* Does the training decrease mental health stigmatizing attitudes and increase cultural identity among trainees?

Participants will complete surveys before and after completing the First Face training, across five time points over the course of two years. Half of the participants will receive the training initially, and half will receive it six months later. Researchers will compare the two groups to examine whether the trainees demonstrate changes in the outcomes of interest compared to the waitlist control group during the first six months, and whether both groups demonstrate sustained changes after the first six months (i.e., once both groups have received training).

DETAILED DESCRIPTION:
For the First Face Training Evaluation study, the researchers will build upon our previous work by evaluating a culturally grounded community mental health training curriculum, First Face for Mental Health. The researchers developed First Face in collaboration with stakeholders from seven Tribal nations to reflect these communities' cultural traditions and values. First Face is a culturally-appropriate community-based mental health training for lay persons and others living and working in Tribal communities that prepares learners to provide assistance to someone having a mental health crisis. By training more individuals in a community to identify, intervene, and connect struggling individuals with the support they need, community culture can be transformed to recognize and address mental health crises.

The overall goal for this First Face Training Evaluation Study (the Research Core component of the Assessing Cultures of Recovery in Tribal Communities Native American Research Centers for Health [NARCH] Center grant issued by NIH) is to evaluate the impact of First Face training both on the trainees and within the Tribal communities as a whole. This Registration covers the evaluation of trainee effects.

The Training Evaluation study will evaluate First Face training using a waitlist control design, implemented in seven tribes, which includes five assessment time points for both initial trainees (n=350) and waitlist controls (n=350). These assessments will measure knowledge about mental health and addiction, as well as the ability and confidence of individuals to respond appropriately to mental health crises.

The researchers will recruit participants from the seven tribes via community-wide announcements and information provided through multiple departments and organizations within each tribe. The Healing Lodge research team and Working Group members will work directly and in person with the tribes to facilitate this recruitment. The researchers will recruit the sample proportional to the size of each tribe (e.g., 30 from the smallest tribe; 280 from the largest). They will assign participants within each tribe as they sign up for the study to either the initial training group or the waitlist control group, based on participant preference, or if no preference, random assignment. To ensure a final recruitment of 700 who are able to attend the trainings, the researchers will attempt to recruit 1,000 initially, allowing a 30% attrition rate for individuals who cannot attend any of the offered training dates.

Multiple trainings of 15-30 individuals will occur separately within each tribe. As shown int he timeline, 350 individuals in the initial training group will receive training and complete a baseline and post-training survey at the time of training. At that same time, the 350 individuals in the waitlist control group will complete an online pre-baseline survey. Six months later, the waitlist control group will undergo training (again, multiple trainings of 15-30 individuals will occur separately within each tribe) and complete baseline and post-training surveys. At the same time, the 350 individuals in the initial training group will complete an online 6 month follow-up survey. Six months later, both groups will complete online surveys - the initial training group will complete their 12-month follow-up and the waitlist control group will complete their 6-month follow-up. Twelve months later, both groups will again complete online surveys -- the initial training group will complete a 24-month follow-up and the waitlist control group will complete an 18-month follow-up.

Note: This study was originally posted as a randomized waitlist control design. We originally intended to block randomize participants within each Tribe to either the initial training group or the waitlist control group as they signed up for the study (and after they had signed the consent form), using a block size of 4. However, across Tribes, it became clear that this type of randomization was not feasible. Organizations within the Tribes where we have gotten permission to advertise and recruit desire for their employees who choose to participate to all take the training at the same time. In many cases, these organizations are providing the time off for their employees to participate. As a result, we are changing our approach to a primarily sequential recruitment procedure. The benefit of the change to randomization is that it allows the Tribal communities to better dictate how they would like to participate in this research and stays true to the principals of Tribal Participatory Research that we follow.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 or older
* Living or working in one of the seven Tribal Nations affiliated with the Healing Lodge of the Seven Nations, including Northwestern United States, including the Coeur d'Alene Tribe, the Confederated Tribes of the Colville Reservation, the Confederated Tribes of the Umatilla Indian Reservation, the Kalispel Tribe of Indians, the Kootenai Tribe of Idaho, the Nez Perce Tribe, and the Spokane Tribe of Indians

Exclusion Criteria:

* Age 13 or younger
* Not living or working in one of the seven Tribal Nations affiliated with the Healing Lodge of the Seven Nations, including Northwestern United States, including the Coeur d'Alene Tribe, the Confederated Tribes of the Colville Reservation, the Confederated Tribes of the Umatilla Indian Reservation, the Kalispel Tribe of Indians, the Kootenai Tribe of Idaho, the Nez Perce Tribe, and the Spokane Tribe of Indians

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mental Health Knowledge | Pre-baseline (6 months before Baseline); Baseline (0 months); Post-training (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  A novel 22-item summed index (possible range from 0 to 22) derived from the First Face Training course to measure knowledge about mental health. Each multiple choice question focuses on a different mental health knowledge item and has one correct answer. Each participant will receive 1 point for each correct answer and 0 points for each incorrect answer. Higher scores indicate a better outcome (i.e., more knowledge about mental health).
Ability to Respond Measured via Situational Judgement Tasks | Pre-baseline (6 months before Baseline); Baseline (0 months); Post-training (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  A novel 7-item measure tapping respondents' ability to respond to and help people experiencing mental health problems (i.e., measured via situational judgment tasks). This measure includes 7 unique vignettes with 5 response options each. Response options are each assigned a value from 1 (least ability to respond) to 5 (greatest ability to respond), and then all are summed to create an overall ability to respond score, with a possible range of 7 to 35. Higher values indicate a better ability to respond to and help people experiencing mental health problems.
Perceived Competence to Respond | Pre-baseline (6 months before Baseline); Baseline (0 months); Post-training (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  A 10-item measure that taps respondents' confidence in their competence to respond to and help people experiencing mental health problems (i.e., Confidence in Recognizing, Intervening and Connecting Individual(s) with Resources Scale; adapted from Talbot et al., 2017). Each response option has a possible range of 1 (Not at all confident) to 5 (Very confident), and a mean will be calculate from all 10 items to yield a scale with a possible range of 1 to 5. Higher values indicate greater perceived competence respond to and help people experiencing mental health problems.
Responsive Actions | Pre-baseline (6 months before Baseline); Baseline (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  Novel measures including 2 items to assess interventions in potential mental health crisis situations in the past 30 days. The first asks "In what ways did you intervene (select all that apply)?", with 4 possible options and an "Other (please specify):" option, and the second asks "What happened after you intervened (select all that apply)?" with 5 possible options and an "Other (please specify):" option. We will report frequencies for these two items at each time point, as these measures are not intended to be summed or averaged into a scale.

SECONDARY OUTCOMES:
Mental Health Stigma Measure 1 | Pre-baseline (6 months before Baseline); Baseline (0 months); Post-training (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  A 22-item scale measuring respondents' stigma toward people experiencing mental health problems (i.e., adapted from the Mental Illness Stigma Scale in Day et al., 2007). Each item has response categories ranging from Completely disagree (coded as 1) to Completely agree (coded as 5), and a mean of all 22 items is calculated to create the scale. The scale has a possible range of 1 to 5, and higher values indicate higher levels of mental health stigma.
Mental Health Stigma Measure 2 | Pre-baseline (6 months before Baseline); Baseline (0 months); Post-training (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  A 21-item scale measuring respondents' stigma toward people experiencing mental health problems (i.e., the Attitudes toward Serious Mental Illness Scale; Watson et al., 2005). Each item has response categories ranging from Completely disagree (coded as 1) to Completely agree (coded as 5), and a mean of all 21 items is calculated to create the scale. The scale has a possible range of 1 to 5, and higher values indicate higher levels of mental health stigma.
Cultural Identity | Pre-baseline (6 months before Baseline); Baseline (0 months); Post-training (0 months); 6 month Follow-up; 12 month Follow-up; 18 month Follow-up; 24 month Follow-up
  A 6-item scale to measure strength of respondents' cultural identity (i.e., adapted from the Multigroup Ethnic Identity Measure - Revised; Phinney & Ong, 2007), which we adapted for this AI/AN population. Each item has 5 responses ranging from Strongly disagree (coded as 1) to Strongly agree (coded as 5), and a mean is calculated from all 6 items to create the scale. The possible range is 1 to 5, and higher values indicate a stronger cultural identity.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E. Nelson, Ph.D., Principal Investigator — Cambridge Health Alliance; Martina Whelshula, Ph.D., Principal Investigator — Healing Lodge of the Seven Nations
Locations (9):
- United States (9):
  - Kootenai Tribe of Idaho, Bonners Ferry, Idaho
  - Nez Perce Tribe, Lapwai, Idaho
  - Coeur d'Alene Tribe, Plummer, Idaho
  - Division on Addiction, Cambridge Health Alliance, Malden, Massachusetts
  - Confederated Tribes of the Umatilla Indian Reservation, Pendleton, Oregon
  - Kalispel Tribe of Indians, Cusick, Washington
  - Confederated Tribes of the Colville Reservation, Nespelem, Washington
  - Healing Lodge of the Seven Nations, Spokane Valley, Washington
  - Spokane Tribe of Indians, Wellpinit, Washington

IPD SHARING:
Plan to Share IPD: No
Each Tribe would need to agree to have their data shared for an IPD plan to be put in place. This has not yet happened, though we will work toward it.

REFERENCES:
- See also: Project Details on NIH RePORT for this funded grant (Assessing Cultures of Recovery in Tribal Communities - Research Core) — https://reporter.nih.gov/search/Fm725t7UakSYoX28Fmgljg/project-details/10437495

DOCUMENTS (3):
  • Informed Consent Form: Informed Consent Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT05998005/ICF_000.pdf
  • Informed Consent Form: Parental Permission Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT05998005/ICF_001.pdf
  • Informed Consent Form: Assent Form Age 14-17 (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT05998005/ICF_002.pdf